CLINICAL TRIAL: NCT04547946
Title: Impact of Melanoma Adjuvant Treatment With Tafinlar® + Mekinist® (Dabrafenib + Trametinib) on Patients Quality of Life (QoL) and Clinical Outcomes in Portuguese Real World Setting
Brief Title: Observational Study for Melanoma Adjuvant Treatment With Tafinlar® + Mekinist® (Dabrafenib + Trametinib)
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CTMT212APT02
Record Dates: First submitted 2020-09-08; First posted 2020-09-14 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Malignant Melanoma
Keywords: Malignant melanoma; Tafinlar; Mekinist; dabrafenib; trametinib; FACT-M questionnaire; generic EQ-5D-3L questionnaire; adjuvant
MeSH Terms: conditions — Melanoma | interventions — dabrafenib; trametinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- dabrafenib + trametinib: Patients administered dabrafenib and trametinib
  Interventions: Drug: dabrafenib + trametinib

INTERVENTIONS:
Drug: dabrafenib + trametinib — There was no treatment allocation. Patients administered adjuvant treatment with combination therapy of Dabrafenib (Tafinlar®) and Trametinib (Mekinist®) by prescription that had started before inclusion of the patient into the study could be enrolled.

SUMMARY:
The primary objective for this non-interventional study was to assess the quality of life of melanoma patients under adjuvant treatment with dabrafenib and trametinib in real world setting in Portugal through disease specific FACT-M questionnaire and generic EQ-5D-3L questionnaire. The secondary study objectives were to assess the usage of adjuvant dabrafenib and trametinib in clinical practice and to evaluate clinical outcomes in patients that started adjuvant treatment with dabrafenib and trametinib. In addition, this study aimed to explore if treatment discontinuation affects clinical outcomes in real-world practice.

DETAILED DESCRIPTION:
The prospective registration of completely resected high-risk stage III melanoma patients treated with dabrafenib and trametinib in the adjuvant setting was planned to be based on collaboration with 8 centers of excellence on melanoma patients treatment, according to their expertise and experience.

Patients were recruited from participating centers in the routine setting. This was done only if the decision about starting treatment with dabrafenib and trametinib had already been made. All patients that complied with the inclusion criteria and that started treatment with dabrafenib+ trametinib during the recruitment period were considered to participate in the study, at investigator discretion.

Health related quality of life had to be assessed by FACT-M and EQ-5D-3L questionnaires after treatment initiation in a quarterly base, according to clinical practice, including the first visit after treatment completion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with complete surgical resection of histologically confirmed AJCC (8th edition) clinical stage III (IIIA, IIIB, IIIC, IIID) melanoma, in whom a decision for adjuvant treatment with dabrafenib and trametinib has been made before entering the study

  * V600E/K mutation-positive cutaneous melanoma
  * Adjuvant treatment with combination therapy of Dabrafenib (Tafinlar®) and Trametinib (Mekinist®) as indicated in the SmPC and by prescription, that has been started before inclusion of the patient into the study;
  * ≥ 18 years of age
  * Written informed consent signed.

Exclusion Criteria:

* Lack of basic demographic (gender, age, age at diagnosis) and staging data (Stage at diagnosis; Breslow index; Clark level; BRAF mutation; BRAF test date; Surgery date).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were recruited from participating centers in the routine setting. This was done only if the decision about starting treatment with darbafenib and trametinib has already been made. All patients that complied with the inclusion criteria and that start treatment with dabrafenib+ trametinib in the participating centers were considered to participate in the study, at investigator discretion.
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2022-06-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in FACT-M score | Baseline, months 3-4, months 6-8, months 9-12, months 12, months 15-16
  Health-related quality of life in melanoma patients defined as the mean difference in FACT-M (Functional Assessment of Cancer Therapy - Melanoma ) score.
  FACT-M is a specific version of FACT questionnaire validated for patients with any stage of melanoma and includes items related to physical, functional, social and emotional well-being, and specific concerns of melanoma patients and melanoma patients undergoing surgery. The FACT-M Total Score (FACT-M TS) ranges from 0 to 172. Higher scores represent a better quality of life.
Change from baseline in EQ-5D-3L score | Baseline, months 3-4, months 6-8, months 9-12, months 12, months 15-16
  Health-related quality of life in melanoma patients defined as the mean difference in EQ-5D-3L score.
  EQ-5D-3L is a descriptive questionnaire comprising five dimensions regarding mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has three response levels of severity: no problems, some problems, extreme problems. The respondent was asked to indicate his/her health state by checking the box next to the most appropriate response level of each of the five dimensions.

SECONDARY OUTCOMES:
Total duration of treatment | months 12
  Total duration of treatment defined as median time on adjuvant treatment (from start to end of treatment/permanent treatment discontinuation).
Proportion of patients on treatment in each visit | Baseline, months 3-4, months 6-8, months 9-12, month 12
  Proportion of patients on treatment in each visit
Rate of permanent study drug discontinuation due to any reason | month 12
  Rate of permanent study drug discontinuation due to any reason.
Rate of permanent drug discontinuation due to pirexia | month 12
  Rate of permanent drug discontinuation due to pirexia over the course of adjuvant treatment.
Rate of permanent drug discontinuation due to AEs | month 12
  Rate of permanent drug discontinuation due to AEs over the course of adjuvant treatment
Reason of treatment discontinuation | month 12
  Reason of treatment discontinuation (death, relapse, AEs, significant change in FACT-M, significant change in EQ-5D-3L , withdrawal of consent, other).
Average dose of dabrafenib and trametinib used during the treatment | month 12
  Average dose of dabrafenib and trametinib used during the treatment, including dose reductions.
Proportion of patients who had dose reduction | month 12
  Percentage of patients with dose reduction during treatment, and in this case, reason for dose reduction
Relapse Free Survival rate | month 12
  RFS (Relapse Free Survival)
distant-metastasis-free survival rate | month 12
  DMFS (distant-metastasis-free survival) rate
Overall Survival rate | month 12
  OS (Overall Survival) rate

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Portugal (2):
  - Novartis Investigative Site, Coimbra, Center
  - Novartis Investigative Site, Porto, North

IPD SHARING:
Plan to Share IPD: No